CLINICAL TRIAL: NCT05835804
Title: Intratumoral Gemcitabine, Paclitaxel, Carboplatine and Intravenous Nivolumab for Locally Recurrence of Head and Neck Cancers
Acronym: NIVOCHIMLOC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI2020_843_0003
Record Dates: First submitted 2023-04-06; First posted 2023-04-28 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Paclitaxel; Carboplatin; Nivolumab
Keywords: Squamous Cell Carcinoma of the Head and Neck; local reccurence of malignant tumor; intrumoral chemotherapy; gemcitabin; paclitaxel; carboplatin; nivolumab
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intratumoral chemotherapy (Experimental)
  Interventions: Drug: GCP intratumoral catheter

INTERVENTIONS:
Drug: GCP intratumoral catheter — After local anaesthesia, intratumoral catheter will be place (one or several depending tumour criteria).The catheter placement could be guided by radiological imaging. Gemcitabine (200mg/l), carboplatin (100mg/l) and paclitaxel (20mg/l) will be each diluted in each in 160ml of NaCl0.9%. GCP will be administered successively for 8hours, at 20ml/h with a total duration of 24hours. The ITC will be done every 28 days for 6 times maximum in case of good response and tolerance. Nivolumab 240 mg IV will be started 1 to 7 days before the first intratumoral infusion and every 15 days, until progression or 2 until years in case of partial response, complete response or stabilization. Evaluation of tumour size will be done by CT-scan, or MRI 2every 2 months and PET-FDG every 3 months.

SUMMARY:
Patients with locally recurrent squamous-cell carcinoma of the head and neck (SCCHN) after Chemotherapy and immunotherapy have a very poor prognosis and limited therapeutic options.

Intratumoral chemotherapy (ITC) with cisplatin and epinephrine in order to increase the local cisplatin retention lead to a 50 % response rate in several studies but was given up due to the poor local tolerance with frequent necrosis of the peritumoral tissues. Gemcitabine, carboplatin and paclitaxel (GCP) are used in advanced SCCHN. These chemotherapies seem to be interesting options for intratumoral infusion: their different effect could lead to avoid chemotherapy resistance with a good tolerance profile, without tissue necrosis profile. The other major option for recurrent SCCHN is immunotherapy by Nivolumab, an anti PD-1 with a 13% mediane response rate. Nevertheless, the failure of this treatment stay unclear, but immunosuppressive action of the tumour is suspected. The presence of tumoral antigen could lead to better response to immunotherapy; association of chemotherapy and immunotherapy seems a promosing association to avoid treatment resistance as cytotoxic release tumoral antigen; it could also be associated to an abscopal effect.

The aim of the study is to evaluate the efficacy of ITC using GCP in LOCAL recurrent SCCHN treated by nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* WHO status : 0, 1 or 2.
* Age > 18ans
* Locally recurrence of a histologically-proven SCCHN after failure of conventional treatments (surgery, radiotherapy, chemotherapy with platinum compounds, cetuximab)
* Nivolumab treatment in second line encouring according to AMM but with insufficient efficacy
* Possible location of the tumour by clinical examination, CT-scan
* Metastases are admitted if there is no vital prognoses threaten and if a clinical benefit is expected by treating local recurrence.
* Neutrophils > 1000/mm3.
* Platelets > 100 000/mm3.
* Blood créatinine < 15 mg/L. Blood bilirubine < 30 mg/L
* Prothrombin rate > 70 %.
* Social insurance
* Informed consent

Exclusion Criteria:

* WHO status : 0, 1 or 2.
* Age > 18ans
* Locally recurrence of a histologically-proven SCCHN after failure of conventional treatments (surgery, radiotherapy, chemotherapy with platinum compounds, cetuximab)
* Nivolumab treatment in second line encouring according to AMM but with insufficient efficacy
* Possible location of the tumour by clinical examination, CT-scan
* Metastases are admitted if there is no vital prognoses threaten and if a clinical benefit is expected by treating local recurrence.
* Neutrophils > 1000/mm3.
* Platelets > 100 000/mm3.
* Blood créatinine < 15 mg/L. Blood bilirubine < 30 mg/L
* Prothrombin rate > 70 %.
* Social insurance
* Informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
local response rate according to RECIST criteria | 3 years
  RECIST is a standard way to measure the response of a tumor to treatment. The criteria to determine whether a tumor disappears, shrinks, are complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD).
  Evaluation of target lesions
  * Complete Response (CR): Disappearance of all target lesions
  * Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD
  * Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started Evaluation of non-target lesions
  * Complete Response (CR): Disappearance of all non-target lesions and no

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No